CLINICAL TRIAL: NCT07306988
Title: Mechanisms of Gut Microbiota in Improving Metabolic Syndrome-Related Parameters Following Helicobacter Pylori Eradication
Brief Title: Eradication of Helicobacter Pylori Improves Metabolic Syndrome Through Modulation of Gut Microbiota.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20250327-12
Record Dates: First submitted 2025-08-29; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-03

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Berberine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VA group (Experimental)
  Interventions: Drug: Vonoprazan-Amoxicillin Dual Therapy
- Probiotics Group (Experimental)
  Interventions: Drug: Vonoprazan-Amoxicillin with Bifidobacterium tetravaccae
- BBR Group (Experimental)
  Interventions: Drug: Vonoprazan-Amoxicillin with Berberine

INTERVENTIONS:
Drug: Vonoprazan-Amoxicillin Dual Therapy — Patients receive oral vonoprazan 20 mg twice daily and amoxicillin 1000 mg three times daily for 14 days. This regimen is a standard dual therapy for Helicobacter pylori eradication.
  Arms: VA group
Drug: Vonoprazan-Amoxicillin with Bifidobacterium tetravaccae — Patients receive oral vonoprazan 20 mg twice daily, amoxicillin 1000 mg three times daily, and Bifidobacterium tetravaccae probiotic tablets (3 tablets three times daily) for 14 days.
  Arms: Probiotics Group
Drug: Vonoprazan-Amoxicillin with Berberine — Patients receive oral vonoprazan 20 mg twice daily, amoxicillin 1000 mg three times daily, and berberine hydrochloride tablets (3 tablets three times daily) for 14 days.
  Arms: BBR Group

SUMMARY:
The Role of Gut Microbiota in the Mechanism of Helicobacter pylori Eradication-Induced Amelioration of Metabolic Syndrome-Related Parameters

Study Sponsor: Nanjing First Hospital Principal Investigator: Dr. Wanli Liu Department: Gastroenterology Study Duration: February 2025 - August 2025

Key Information for Patients and Families

1. What is this study about? This study aims to understand how treating a common stomach infection caused by Helicobacter pylori (Hp) might improve metabolic health issues like high blood sugar, cholesterol problems, or obesity (collectively called metabolic syndrome). Specifically, it explores whether adding probiotics (good bacteria) or a natural compound called berberine (BBR) to standard Hp treatment can enhance these benefits by improving gut bacteria balance.
2. Who can participate? Patients: Adults aged 18-65 with both Helicobacter pylori infection (confirmed by a breath test) and newly diagnosed metabolic syndrome (based on waist size, blood sugar, cholesterol, or blood pressure).

   Healthy Volunteers: Adults aged 18-65 with no Hp infection and normal metabolic health (to compare results).

   Exclusions:

   Allergy to study medications (e.g., penicillin).

   Previous Hp treatment, recent antibiotic/steroid use, pregnancy, or serious medical conditions (e.g., liver/kidney disease).
3. What will participants do?

   Treatment Groups:

   Group A: Take two medications (vonoprazan + amoxicillin) for 14 days.

   Group B: Take the two medications + probiotics (Bifidobacterium tablets).

   Group C: Take the two medications + berberine (a plant-based supplement).

   Tests:

   Before treatment: Breath test, blood tests (blood sugar, cholesterol, inflammation markers), stool sample analysis (gut bacteria), and body measurements (weight, waist size).

   After treatment (1 month): Repeat tests to check Hp eradication and metabolic improvements.
4. Possible Benefits and Risks

   Benefits:

   Free Hp treatment and metabolic health monitoring.

   Potential improvement in blood sugar, cholesterol, or weight.

   Contribution to future treatments for metabolic syndrome.

   Risks:

   Mild side effects (e.g., nausea, diarrhea, stomach pain) from medications.

   Discomfort from blood draws or stool sample collection.
5. How are participants protected? All treatments are FDA-approved or widely used in clinical practice.

Ethical review ensures participant safety.

You can withdraw at any time without affecting your regular care.

Information for Health Care Providers

1. Study Design Type: Prospective, single-center, open-label, randomized controlled trial.

   Population: 140 participants (120 Hp+ patients with metabolic syndrome; 20 Hp- healthy controls).

   Intervention:

   Group A: Vonoprazan (20 mg bid) + amoxicillin (1 g tid) for 14 days.

   Group B: Group A + Bifidobacterium tetragenous probiotic (3 tablets tid).

   Group C: Group A + berberine (3 tablets tid).

   Primary Outcomes:

   Hp eradication rate (confirmed by urea breath test).

   Changes in metabolic parameters (fasting glucose, HbA1c, lipid profile).

   Gut microbiota composition (16S rRNA sequencing).

   Secondary Outcomes:

   Multi-omics analysis (inflammation markers, endotoxins, short-chain fatty acids, bile acids).
2. Scientific Rationale Hp and Metabolic Syndrome: Epidemiological evidence links Hp infection to metabolic dysfunction, possibly via chronic inflammation. Eradication may partially reverse insulin resistance and dyslipidemia.

   Gut Microbiota as Mediator: Hp eradication alters gut microbiota, which regulates metabolic homeostasis through metabolites (e.g., SCFAs), bile acid metabolism, and inflammatory pathways. Probiotics/BBR may enhance these effects.
3. Methodology Randomization: Block randomization (block size = 4) using SAS 9.4.

   Assessments:

   Metabolic Parameters: Fasting glucose, HbA1c, lipid profile, BMI.

   Microbiome: 16S rRNA sequencing (α/β diversity, taxa abundance).

   Multi-omics: ELISA (TNF-α, IL-6), GC-MS (SCFAs), UPLC-MS (bile acids).

   Statistical Analysis:

   Microbiome: QIIME2, LEfSe, PICRUSt2.

   Multi-omics: limma, SparCC, sPLS-DA.

   Clinical data: ANOVA, χ² tests (SPSS v25.0).
4. Clinical Implications Clarify whether probiotics or BBR add value to Hp eradication in improving metabolic health.

Identify gut microbiota-driven mechanisms linking Hp eradication to metabolic benefits.

Resources for Participants

Study Flowchart:

Screening: Breath test, blood/stool tests (1 week).

Treatment: 14 days of medication.

Follow-up: Repeat tests at 1 month.

Contact Information:

Dr. Wanli Liu: +86-18951670222

Nanjing First Hospital Gastroenterology Department.

FAQ Sheet:

Can I take my regular medications? Yes, unless they interfere with Hp treatment (e.g., PPIs).

What if I miss a dose? Contact the study team immediately.

Ethical Compliance Approved by the Institutional Review Board of Nanjing First Hospital.

Complies with the Declaration of Helsinki and China's ethical guidelines.

Informed consent required for participation.

ELIGIBILITY:
Inclusion Criteria:

* For H. pylori-naïve infected patients with newly diagnosed metabolic syndrome (MS):

  1. Aged 18-65 years;
  2. Confirmed H. pylori-positive status by urea breath test (UBT), with no prior eradication therapy;
  3. Newly diagnosed MS according to the Chinese Diabetes Society (CDS, 2004 Chinese criteria) ;
  4. Voluntarily join the trial and sign informed consent.
* For H. pylori-negative healthy controls with normal metabolism:

  1. Aged 18-65 years;
  2. Confirmed H. pylori-negative status by UBT;
  3. Normal metabolic parameters (e.g., blood glucose, lipid profile, blood pressure) without MS;
  4. Voluntarily join the trial and sign informed consent.

Exclusion Criteria:

1. Hypersensitivity to study drugs (e.g., penicillin, amoxicillin, vonoprazan);
2. Active peptic ulcer confirmed by endoscopy;
3. Prior history of H. pylori eradication therapy;
4. Use of medications for metabolic regulation (e.g., hypoglycemic agents, lipid-lowering drugs, weight-loss drugs)
5. Recent use of antibiotics or bismuth (within 4 weeks) or H2-receptor antagonists/PPIs (within 2 weeks) before enrollment;
6. Current use of corticosteroids, NSAIDs, or anticoagulants;
7. History of esophageal or gastric surgery;
8. Pregnant or breastfeeding women;
9. Severe comorbidities (e.g., hepatic, cardiovascular, pulmonary, renal diseases, inflammatory bowel disease);
10. Chronic alcohol abuse (>40 g/day for men, >20 g/day for women);
11. Malignancies (e.g., gastric mucosa-associated lymphoid tissue [MALT] lymphoma).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori Eradication Rate | Post-treatment follow-up at 1 month
Change in Serum Triglycerides | Baseline and 1 month post-treatment.
Change in HDL Cholesterol | Baseline and 1 month post-treatment.
Change in Blood Pressure | Baseline and 1 month post-treatment.
Change in Waist Circumference | Baseline and 1 month post-treatment.
Change in Fasting Plasma Glucose | Baseline and 1 month post-treatment.

SECONDARY OUTCOMES:
Change in gut microbiota alpha-diversity, assessed by 16S rRNA gene sequencing | Baseline and 1 month post-treatment.
Change in gut microbiota beta-diversity, assessed by 16S rRNA gene sequencing | Baseline and 1 month post-treatment.
Identification of differentially abundant bacterial taxa (Genus level), assessed by 16S rRNA gene sequencing and statistical modeling (e.g., LEfSe or DESeq2) | Baseline and 1 month post-treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No